CLINICAL TRIAL: NCT04664387
Title: EARLY Assessment of Somatic Symptom Disorder in Patients With MYOcardial Bridge by Somatic Symptom Scale China (SSS-CN) (EARLY-MYO-SSS-CN-Ⅱ)
Brief Title: Somatic Symptom Disorders in Patients With Myocardial Bridge
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SSSCN202010
Record Dates: First submitted 2020-12-06; First posted 2020-12-11 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2020-10

CONDITIONS: Myocardial Bridge; Somatic Symptom Disorder
Keywords: myocardial bridge; somatic symptom disorder; SSS-CN
MeSH Terms: conditions — Myocardial Bridging | interventions — Coronary Angiography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with myocardial bridge: patients who underwent coronary angiography and was diagnosed as myocardial bridge
  Interventions: Diagnostic Test: coronary angiography
- patients without myocardial bridge: patients who underwent coronary angiography and was diagnosed as without myocardial bridge
  Interventions: Diagnostic Test: coronary angiography

INTERVENTIONS:
Diagnostic Test: coronary angiography — A coronary angiography is a test to find out if there is stenosis in coronary artery.

SUMMARY:
The purpose of this study was to investigate the prevalence of physical and mental disorder in the population of patients with myocardial bridge and to describe the relationship between clinical features and the occurrence of somatic disorder.

DETAILED DESCRIPTION:
Myocardial bridge (MB), a congenital cardiac anomaly, is an unignored contribution to chest pain. Patients with MB often complain about chest discomfort more serious than the degree of vessel compression. The symptoms are also often inconsistence with the degree of coronary stenosis. Reports suggested that patients with MB may companioned with depression and anxiety. Moreover, patients with MB often have other systemic complaints including stomach pain, pain on the back, ear blockage, et al. Investigators assume that somatic symptom disorder (SSD) may play a part in aggregating the severity of symptoms. In order to screen SSD, investigators previously developed the Somatic Symptom Scale-China (SSS-CN) questionnaire. It is a somatic and psychological symptom scale which was developed based on the DSM-5 to assess a combination of psychological, behavioral and somatic symptoms. It is designed to assess the presence and severity of the symptoms. Investigators have validated its reliability and validity in a previous study. The purpose of this study was to investigate the prevalence of physical and mental disorder in the population of patients with MB and to describe the relationship between clinical features and the occurrence of somatic disorder.

ELIGIBILITY:
Inclusion Criteria:

* cardiology inpatients with the age older than 18, complained with chest discomfort and was suspected with coronary artery disease.
* undertook Somatic Symptom Scale-China (SSS-CN) questionnaire, Patient Health Questionnaire-9 (PHQ-9) and Generalized Anxiety Disorder-7 (GAD-7) questionnaires.
* underwent cardiac angiography.
* agree to participate.

Exclusion Criteria:

* patients who are in emergency or unconsciousness.
* patients who refuse to participate or with unfinished questionnaire.
* the questionnaires were undertook after the angiography.
* patients who have previously been confirmed to have mental disorders, mental retardation or dementia, cannot finish questionnaires
* patients who currently take anti-anxiety or anti-depression agents.
* patients who have been confirmed to have heart diseases other than coronary vascular disease.
* patients who have been previously confirmed to have other physical diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive suspected CAD inpatients from Renji cardiology department.
Sampling Method: Non-Probability Sample
Enrollment: 1357 (Actual)
Dates: Start 2016-10-30 (Actual); Primary Completion 2020-05-08 (Actual); Study Completion 2020-05-08 (Actual)

PRIMARY OUTCOMES:
the score of Somatic Symptom Scale-China (SSS-CN) | within 24 hours before the coronary angiography.
  to compare the score of Somatic Symptom Scale-China questionnaire between patients with and without myocardial bridge. SSS-CN is a self-administered questionnaire with 20 items and scoring 1, 2, 3, 4 to each item. The total score is from 20 to 80. The higher the score is, the higher frequency that the symptoms presented.

CONTACTS AND LOCATIONS:
Overall Officials: Meng Jiang, MD, Study Chair — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, China